CLINICAL TRIAL: NCT06035328
Title: Comparison Efficacy Between Two Different Frequency of Maintenance Dose-oral Immunotherapy for Children With Wheat Allergy
Brief Title: Comparison Efficacy Between Two Different Frequency of Maintenance Dose Oral Immunotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 069/2566(IRB3)
Record Dates: First submitted 2023-04-18; First posted 2023-09-13 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Wheat Hypersensitivity; Immunotherapy
Keywords: Wheat Hypersensitivity; Immunotherapy; Short term unresponsiveness
MeSH Terms: conditions — Wheat Hypersensitivity | interventions — Flour

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Four per week (Experimental): Case wheat allergy that on four times/week dose during one year maintenance phase of wheat OIT
  Interventions: Other: Wheat (Four times per week)
- Once daily (No Intervention): Case wheat allergy that on once daily dose during one year maintenance phase of wheat OIT

INTERVENTIONS:
Other: Wheat (Four times per week) — Case wheat allergy that on four times/week dose during one year maintenance phase of wheat OIT
  Arms: Four per week

SUMMARY:
Oral immunotherapy(OIT) is effective in desensitized food allergy. OIT protocols are not standardized, and a wide heterogeneity exists in the literature . So the purpose of our study is to compare short term unresponsiveness rate between once daily dose and four times/week dose during one year maintenance phase of wheat OIT

DETAILED DESCRIPTION:
All subject in this study were patients with history of IgE mediated wheat allergy and positive OFC test. All of them received wheat OIT and reached target maintenance dose of wheat OIT.

The primary outcome was to compare short term unresponsiveness rate between once daily dose and four times/week dose during one year maintenance phase of wheat OIT. Other outcomes were collected during the projected such as blood and skin examination for immunologic parameter, changing in Body weight, WA, WH and BMI, compliance, adverse reactions, rates of medication used during OIT and quality of life

ELIGIBILITY:
Inclusion Criteria:

* Age 5-18 years old
* Children aged 5-18 years with history of IgE mediated wheat allergy and positive OFC test
* Reach target maintenance dose of wheat OIT and ongoing to maintenance phase of wheat OIT

Exclusion Criteria:

* Patient with low dose OIT protocol
* Patients with uncontrolled atopic dermatitis, uncontrolled asthma, or any chronic disease;
* Patients who had been treated with some other immunotherapy (eg, SLIT, another OIT) or biologic therapy (eg, Omalizumab)
* Patients with a developmental problem or mental disorder
* Active eosinophilic gastrointestinal disease in the past 2 years
* Use of b-blockers (oral), angiotensin-converting enzyme inhibitors, angiotensin-receptor blockers, or calcium-channel blockers
* Pregnancy or lactation
* Patient who could not visit clinic as protocol

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2027-03-22 (Estimated); Study Completion 2027-03-22 (Estimated)

PRIMARY OUTCOMES:
Short term unresponsiveness rate | 13 months
  Short term unresponsiveness rate between once daily dose and four times/week dose .during maintenance phase of wheat OIT.
  Short term unresponsiveness means patients who pass the oral food challenge test after stopping oral immunotherapy for a short period

SECONDARY OUTCOMES:
Specific IgE to wheat | 13 months
  Specific IgE to wheat
Specific IgG4 to wheat | 13 months
  Specific IgG4 to wheat
Changing in Body weight | 13 months
  Changing in Body weight in kilograms
Compliance | 12 months
  Compliance of wheat ingestion (group A: every day, groupB: 4 days/weeks). Compliance can be calculated by dividing the number of days on which wheat is actually ingested by the total number of days prescribed for wheat consumption.
Adverse reactions | 13 months
  Adverse reaction during treatment will be recorded by using WAO systemic allergic reaction grading system
Quality of life by using FAQLQ-PF | 13 months
  Quality of life before and after enrollment by using FAQLQ-PF

CONTACTS AND LOCATIONS:
Overall Officials: Punchama Pacharn, MD, Principal Investigator — Mahidol University, Siriraj Hospital,Thailand
Locations (1):
- Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pajno GB, Fernandez-Rivas M, Arasi S, Roberts G, Akdis CA, Alvaro-Lozano M, Beyer K, Bindslev-Jensen C, Burks W, Ebisawa M, Eigenmann P, Knol E, Nadeau KC, Poulsen LK, van Ree R, Santos AF, du Toit G, Dhami S, Nurmatov U, Boloh Y, Makela M, O'Mahony L, Papadopoulos N, Sackesen C, Agache I, Angier E, Halken S, Jutel M, Lau S, Pfaar O, Ryan D, Sturm G, Varga EM, van Wijk RG, Sheikh A, Muraro A; EAACI Allergen Immunotherapy Guidelines Group. EAACI Guidelines on allergen immunotherapy: IgE-mediated food allergy. Allergy. 2018 Apr;73(4):799-815. doi: 10.1111/all.13319. Epub 2017 Dec 5. PMID 29205393